CLINICAL TRIAL: NCT01953185
Title: MANUAL DIAPHRAGM RELEASE TECHNIQUE INCREASES TIDAL VOLUME AND UPPER RIB CAGE CONTRIBUTION DURING QUIET BREATHING IN ELDERLY: A RANDOMIZED CONTROLLED TRIAL
Brief Title: MANUAL DIAPHRAGM RELEASE TECHNIQUE INCREASES TIDAL VOLUME IN ELDERLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniella Cunha Brandao (Other)
Responsible Party: Sponsor-Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: taciano01
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: elderly; subjects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual diaphragm release technique (Experimental)
  Interventions: Other: The manual diaphragm release technique
- Control group (Sham Comparator)
  Interventions: Other: Sham manual diaphragm release technique

INTERVENTIONS:
Other: Sham manual diaphragm release technique — For this group, light touch at the same anatomical points was done without exerting pressure or traction. Positioning and duration were identical to the IG to perform the sham protocol (Licciardone & Russo, 2006).
  Arms: Control group
Other: The manual diaphragm release technique — To perform the technique the volunteer was placed in supine position with limbs relaxed. Positioned behind the head of the volunteer, the therapist performed manual contact (pisiform, ulnar edge and the last three fingers) with the underside of the costal cartilage of the 7th, 8th, 9th and 10th rib, and guiding forearms toward the shoulders of the corresponding side. In the inspiratory phase, the therapist gently pulled the points of contact with both hands, in the direction of the head, yet slightly lateral, accompanying the elevation movement of the ribs. During exhalation, the therapist deepened contact toward the inner costal, maintaining resistance throughout the inspiratory phase. In the breaths following, the therapist sought to gain traction and smooth increase in the deepening of contacts. This maneuver was performed in two sets of ten deep breaths, with a one minute interval between them.
  Arms: Manual diaphragm release technique

SUMMARY:
Question: Does manual diaphragm release change kinematics and respiratory function of elderly subjects? Design: Randomized controlled trial with concealed allocation and double-blinding.

Participants: 17 volunteers over 60 years old randomized into two groups: 09 in the Control Group (CG) and 08 in the Intervention Group (IG).

Intervention: The manual diaphragm release technique was used on the IG, in two sets of ten deep breaths, with a one minute interval between them. The CG underwent a sham protocol (light touch), with same sets and time of interval.

Outcome measures: The groups were evaluated using spirometry, manovacuometry and optoelectronic plethysmography (OEP), in that order, before and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years of age;
* a body mass index (BMI) below 30 kg/m2
* non-smokers, self-declared sedentary;
* presenting a forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) greater than or equal to 80% of predicted;
* the ratio between these variables (FEV1/FVC) greater than 70% in spirometry

Exclusion Criteria:

* Showed the inability to understand verbal commands in the evaluation.

Ages: 60 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Compartmental chest wall volume | 1 day

SECONDARY OUTCOMES:
Pulmonary function | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Taciano Rocha, Msc, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Aliverti A, Pedotti A. Opto-electronic plethysmography. Monaldi Arch Chest Dis. 2003 Jan-Mar;59(1):12-6. PMID 14533277
- [Result] De Troyer A. Respiratory effect of the lower rib displacement produced by the diaphragm. J Appl Physiol (1985). 2012 Feb;112(4):529-34. doi: 10.1152/japplphysiol.01067.2011. Epub 2011 Dec 1. PMID 22134697